CLINICAL TRIAL: NCT01024465
Title: ReShape Intragastric Balloon for the Treatment of Obesity
Acronym: ITALYIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReShape Lifesciences (Industry)
Collaborators: Regional Hospital. Viale Rodolfi 37. 36100 Vicenza. ITALY (Unknown); Casa di Cura Solatrix. Via Bellini 11. 38068 Rovereto. ITALY (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-1
Record Dates: First submitted 2009-11-25; First posted 2009-12-02 (Estimated); Results first posted 2015-09-11 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: obesity; intragastric balloon
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReShape Duo Balloon (Experimental): Patients seeking weight loss with a starting BMI in the 30-40 range, received the ReShape Duo Balloon
  Interventions: Device: ReShape Duo Balloon

INTERVENTIONS:
Device: ReShape Duo Balloon — ReShape Duo Balloon

SUMMARY:
A prospective, non-randomized, open-label, multi-center study designed to implant up to twenty-six (26) CE-marked ReShape™ Balloons in twenty-six (26) patients with body mass index (BMI) 30-40 to assess the effectiveness of the device. The RIB devices will be used within their labeled indications and as per their instructions for use. Enrolled patients will be followed for seven months. The patient will be prescribed a controlled diet, exercise and counseling. One group of 26 patients will receive treatment as follows: Placement, inflate to 900 cc, remove at 180 days, follow-up 30 days post removal (endoscopic video capture of placement and removal required).

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female between the ages of 20 and 60 years of age.
* The patient presents with a Body Mass Index (BMI) 30-40 kg/m2.
* The patient is geographically stable and willing to return to the implant center for follow-up visits.
* The patient has been adequately informed of risks and requirements and consents to his/her participation in the post market clinical study.

Exclusion Criteria:

* The patient presents with 20 years > Age > 60 years.
* The patient has a progressive disease, which in the Investigator's experience produces an unacceptable increased risk to the patient, or results in a life expectancy of less than 12 months.
* The patient is a pregnant or lactating female.
* The patient presents with a 30 kg/m2 > BMI > 40 kg/m2.
* The patient has had previous abdominal surgery.
* The patient has digestive tract disorders such as active peptic ulcers, bleeding disorders, esophageal varices, Crohn's disease.
* The patient presents with psychiatric disorders.
* The patient is participating in concomitant research studies of investigational products that would interfere with this study.
* The patient has inability to return for follow-up assessments.
* The patient is an alcohol or drug abuser.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Mooney, Study Director — ReShape Medical
Locations (2):
- Italy (2):
  - Casa di Cura Solatrix, Rovereto
  - Regional Hospital, Vicenza

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ReShape Duo Balloon
Started | 26
Completed | 23
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants were enrolled who met the study's inclusion/exclusion criteria.
Arm/Group | ReShape Duo Balloon
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Weight Loss
Description: Mean weight loss in kilograms compared with the baseline value through 6 months of study follow up.
Time Frame: baseline to 180 days
Population: Subjects with a weight recorded at 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | ReShape Duo Balloon
Number analyzed (Participants) | 22
kg | -9.4 (6.3)

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | ReShape Duo Balloon
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 16/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ReShape Duo Balloon (N=26)
nausea/vomiting after discharge (Gastrointestinal disorders) | 4
gastric bloating (Gastrointestinal disorders) | 4
epigastric pain (Gastrointestinal disorders) | 3
GERD (Gastrointestinal disorders) | 3
ulcer at removal (Gastrointestinal disorders) | 3
diarrhea (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
No limitations nor caveats apply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon study conclusion, the PI has the right to use the study data for educational purposes, scientific conferences and publications. The sponsor will have a period of 15 days (for abstracts) and 30 days (for scientific publications) to review the proposal for disclosure / publication for the sole purpose of protecting any confidential information. If such disclosure contains Confidential Information, the PI agrees to remove such Confidential Information.